CLINICAL TRIAL: NCT01131845
Title: An Evaluation of the Pharmacokinetics and Safety of a Single Dose of UT-15C SR (Treprostinil Diethanolamine) in Subjects With Renal Impairment.
Brief Title: The Effect of Renal Impairment on the Pharmacokinetics of Oral Treprostinil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-120
Record Dates: First submitted 2010-05-10; First posted 2010-05-27 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Pulmonary Arterial Hypertension; Renal Dysfunction
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Renal Insufficiency | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treprostinil diethanolamine (Experimental)
  Interventions: Drug: UT-15C SR (treprostinil diethanolamine)

INTERVENTIONS:
Drug: UT-15C SR (treprostinil diethanolamine) — Single dose, 1 mg UT-15C SR

SUMMARY:
This is a single-center, open-label, single-dose evaluation of 1 mg UT-15C SR pharmacokinetics, safety, and tolerability in subjects with normal, mild, moderate and end stage renal disease (ESRD; on dialysis).

Subjects in the ESRD group will receive 2 doses of UT-15C SR, separated by 14 days. One dose will be given 4 hours prior to dialysis, the other dose will be given at the end of dialysis.

Pharmacokinetic samples will be taken immediately prior to dosing and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 24, 30, 36, 42 and 48 hours post dose. Additionally, subjects with ESRD will have a sample taken at 60 hrs post dose.

ELIGIBILITY:
Male and female volunteers with ESRD (requiring dialysis), moderate (creatinine clearance; CrCL = 30-50 mL/min), mild (CrCL = 50-80 mL/min) and normal renal function (control group; (CrCL >80 mL/min)) may be enrolled. Eligible subject will be 18-79 years of age with a BMI between 18 - 40 kg/m2 and not taking chronic nonsteroidal antiinflammatory drugs (NSAIDs)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Treprostinil pharmacokinetics in volunteers with varying degrees of renal function following a single oral dose of a 1 mg treprostinil diethanolamine sustained release. | 48hrs post dose (60 hours for ESRD)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marbury, MD, Principal Investigator — Orlando Clincal Reserach Center
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States